CLINICAL TRIAL: NCT03083262
Title: Retrospective Chart Review to Investigate an Association Between Vulvovaginal Atrophy and High Tone Pelvic Floor Dysfunction (HTPFD)
Brief Title: High Tone Pelvic Floor Dysfunction
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Becky Lynn, MD, Principal Investigator, St. Louis University
Other Study IDs: 27975
Record Dates: First submitted 2017-03-03; First posted 2017-03-17 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Vulvovaginal Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — None, there is no intervention

SUMMARY:
Dyspareunia, or painful intercourse, is one of the most commonly reported complaints in postmenopausal women. One common cause of dyspareunia is vaginal atrophy (VVA), which occurs in >50% of postmenopausal women. At the time of menopause, a lack of estrogen thins the vaginal mucosa and lessons lubrication, making sex painful. Some women with vaginal atrophy will also have high tone pelvic floor dysfunction (HTPFD) (also known as levator spasm). Successful treatment of the sexual pain requires treatment of both vaginal atrophy and HTPFD.

How often vaginal atrophy and HTPFD coexist has not been studied. In fact, the prevalence of HTPFD is unknown. This is most likely due to the fact that many clinicians are unaware of its existence or how to diagnose or treat it. Also, sexual symptoms tend to be underreported due to embarrassment or hesitation to seek care. HTPFD frequently coexists with other conditions that cause pain like vaginal atrophy, endometriosis or interstitial cystitis. Treatment includes treating both conditions. If only one is treated, then sexual pain is likely to continue. There are several available treatments for HTPFD that have been studied including physical therapy, botox and intravaginal diazepam.

This is an area where clinicians may be under treating a condition and limiting the possibility of restoring normal sexual function to many women. Treating only vaginal atrophy without appropriate evaluation and treatment of HTPFD leaves a cohort of women still struggling with sexual pain. With a better understanding of the relationship between HTPFD and vaginal atrophy, the investigators hope to bring awareness concerning the importance of treating both in restoring normal sexual function.

DETAILED DESCRIPTION:
This is a retrospective chart review that will be performed to identify all female patients in the electronic medical records with a diagnosis of vulvovaginal atrophy (VVA).

The records of these patients with VVA will be examined for demographics, symptoms, answers to standardized questionnaires ( e.g. Female Sexual Function Index - FSFI - that is routinely assessed during clinical evaluation), work-up, diagnosis, and/or treatment of high tone pelvic floor dysfunction (HTPFD). Symptoms of HTPFD include but are not limited to pelvic pressure or pain, and dyspareunia. These data will then undergo statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of vulvovaginal atrophy (VVA)

Exclusion Criteria:

* not meeting the inclusion criteria

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: >/= 18 -90 years of age female any ethnic background
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
vulvovaginal atrophy | 3 months
  Charts reviewed for HTPFD

CONTACTS AND LOCATIONS:
Overall Officials: Becky K Lynn, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No